CLINICAL TRIAL: NCT03420235
Title: Home Monitoring in Idiopathic Pulmonary Fibrosis; Improving Use of Anti-fibrotic Medication and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: OLVG (Network); St. Antonius Hospital (Other); Zuyderland Medical Centre (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Dr. M.S. Wijsenbeek, pulmonologist, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL62925.078.17
Record Dates: First submitted 2017-12-20; First posted 2018-02-05 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: quality of life; eHealth; patient-reported outcomes; home spirometry; cost-effectiveness; home monitoring
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized clinical multi-center study to evaluate the effect of home monitoring on disease-specific HRQOL, (appropriate) medication use and other patient-relevant outcomes in patients with IPF treated with anti-fibrotic drugs. Patients with IPF about to start on anti-fibrotic medication will be randomly assigned to receive either the home monitoring program integrated with standard care or standard care alone after informed consent. Patient will be stratified for study center and medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group will receive standard care alone.
- Home monitoring group (Experimental): Intervention will consist of a home monitoring program added to standard care.
  Interventions: Other: Home monitoring program

INTERVENTIONS:
Other: Home monitoring program — The home monitoring program consists of 1) the use of an interactive internet tool to coach patients and enhance self-management 2) home-based pulmonary function testing with a handheld spirometer and 3) recording of patient-reported outcomes (PROs).
  Arms: Home monitoring group

SUMMARY:
In this study it will be investigate whether a home monitoring program improves disease-specific health-related quality of life (HRQOL) for patients with idiopathic pulmonary fibrosis (IPF) through appropriate medication use and subsequently results in better objective and subjective outcomes.

DETAILED DESCRIPTION:
IPF is a chronic disease with progressive scarring of the lung tissue (fibrosis), resulting in a poor prognosis and a devastating impact on the lives of patients and their families. Progressive shortness of breath, cough and fatigue are major factors influencing health-related quality of life (HRQOL) in patients with IPF. Recently two anti-fibrotic drugs became available that slow down disease progression. The availability of effective drugs for this devastating disease has importantly changed daily care and research in IPF. Currently, one of the major challenges in daily IPF care is the evaluation of how individual patients objectively and subjectively experience treatment and benefit from treatment. The use of information communication technology in health care, also named e-health, is a promising solution to improve the quality of care. E-health allows remote exchange of data between patients and health care professionals which enables monitoring, research and management of long term conditions. Also communication between patients and physicians, and physicians mutually, becomes more accessible. This creates an opportunity for earlier intervention by health care professionals, which may prevent a hospital admission. This might improve quality of life and reduce costs. Patients easily get access to up-to-date and tailored information, in an interactive way. By providing these tools, patients may better understand their health conditions and become actively involved in management of their own health care, which may lead to a better health status. An 'internet tool' for patients with IPF have been developed, providing information and enabling them to keep track of their own symptoms, HRQOL scores, medication use and lung function results.

In this study it will be investigated whether a home monitoring program improves disease-specific HRQOL for IPF patients through appropriate medication use and subsequently results in better objective and subjective outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of IPF according to the ATS 2011 criteria and about to start on anti-fibrotic treatment (either nintedanib or pirfenidone)

Exclusion Criteria:

* Not able to speak, read or write in Dutch
* No access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Difference in the change in total score of King's brief Interstitial Lung Disease Health Status (K-BILD) questionnaire between the home monitoring group and the standard care group | 24 weeks after inclusion
  Change in HRQOL assessed by the K-BILD, between control group and home monitoring group at the end of the study. The K-BILD is a 15-item self-administered questionnaire on a 7-point response scale. It has three domains: breathlessness and activities, psychological and chest symptoms.The domain and total score ranges are 0-100, with the higher scores corresponding with better HRQL.

SECONDARY OUTCOMES:
Difference in the change in total score of King's brief Interstitial Lung Disease Health Status (K-BILD) questionnaire between the home monitoring group and the standard care group | 12 weeks after inclusion
  Change in HRQOL assessed by the K-BILD, between control group and home monitoring group. The K-BILD is a 15-item self-administered questionnaire on a 7-point response scale. It has three domains: breathlessness and activities, psychological and chest symptoms.The domain and total score ranges are 0-100, with the higher scores corresponding with better HRQL.
Patient-reported outcome (PRO) scores (GRC) | 12 weeks after inclusion
  Patients will fill in the Global Rating of Change (GRC) which measures whether QoL has improved or deteriorated over a certain period of time, with scores range from -7 to +7, with positive scores corresponding with improvement in QoL
Patient-reported outcome (PRO) scores (EQ5D) | 12 weeks after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
Patient-reported outcome (PRO) scores (HADS) | 12 weeks after inclusion
  Patients will complete the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire with 7 questions in the domain anxiety and 7 questions in the domain depression on a 0-3 Likert scale. Higher values represent higher anxiety and depression levels, with a maximum of 21 point in both domains. There is a cut-off score of 8/21 for anxiety and depression.
Patient-reported outcome (PRO) scores (HADS) | 24 weeks after inclusion
  Patients will complete the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire with 7 questions in the domain anxiety and 7 questions in the domain depression on a 0-3 Likert scale. Higher values represent higher anxiety and depression levels, with a maximum of 21 point in both domains. There is a cut-off score of 8/21 for anxiety and depression.
Patient-reported outcome (PRO) scores (EQ5D) | 24 weeks after inclusion
  Patients will complete the EQ-5D-5L questionnaire, a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
Patient-reported outcome (PRO) scores (GRC) | 24 weeks after inclusion
  Patients will complete the Global Rating of Change (GRC) which measures whether QoL has improved or deteriorated over a certain period of time, with scores range from -7 to +7, with positive scores corresponding with improvement in QoL.
Patient expectations and satisfaction with medication (PESaM scores) | Baseline and 12 weeks after inclusion
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 12 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient expectations and satisfaction with medication (PESaM scores) | Baseline and 24 weeks after inclusion
  Correlation between patient expectations with medication and consecutive experiences measured with the PESaM questionnaire which assess patient expectations at baseline in an 11-item questionnaire and patient experiences and side-effects with medication after 24 weeks in a 26-item questionnaire on a 0-4 Likert scale. For each question it is different whether a higher score represents better or worse outcomes.
Patient satisfaction with medication (PESaM scores) | 24 weeks after inclusion
  Overall patient satisfaction with medication after 24 weeks resulting from the 26-item PESaM questionnaire. For each question it is different whether a higher score represents better or worse outcomes
Patient satisfaction with the care process | 24 weeks after inclusion
  Evaluation and satisfaction questionnaire at the end of the study. 10-item questionnaire with answers on a scale from -5 to 5, with higher scores corresponding with higher satisfaction
Number of patients who discontinue use of medication, pills used and pills wasted | 24 weeks after inclusion
  Every week patients register whether they missed pills (and the amount of pills wasted). Discontinuation or switch of medication is registered both by patients and researchers.
Amount of contacts with healthcare providers and number of visits per patient | 24 weeks after inclusion
  During the study patients register their contacts with healthcare providers (hospital visits, general practitioner visits, physiotherapist, dietician, psychologist), after 24 weeks the amount of contacts will be assessed
FVC decline | 12 weeks after inclusion
  FVC decline measured by hospital-based spirometry and daily home spirometry
FVC decline | 24 weeks after inclusion
  FVC decline measured by hospital-based spirometry and daily home spirometry
Personal goal of patient defined at start of study | 24 weeks after inclusion
  Change in score of personal goal. Patients define a personal goal at the start of the study and they score on a scale from 0 -10 how far they have reached their goal

OTHER OUTCOMES:
Home monitoring values of FVC compared to in hospital values of lung function | 12 weeks after inclusion
  Home monitoring values compared to in hospital values of lung function
Home monitoring values of FVC compared to in hospital values of lung function | 24 weeks after inclusion
  Home monitoring values compared to in hospital values of lung function
Correlation between FVC measurements and K-BILD | 12 weeks after inclusion
  Correlation between FVC and K-BILD. The K-BILD is a 15-item self-administered questionnaire on a 7-point response scale. It has three domains: breathlessness and activities, psychological and chest symptoms.The domain and total score ranges are 0-100, with the higher scores corresponding with better HRQL.
Correlation between FVC measurements and K-BILD | 24 weeks after inclusion
  Correlation between FVC and K-BILD. The K-BILD is a 15-item self-administered questionnaire on a 7-point response scale. It has three domains: breathlessness and activities, psychological and chest symptoms.The domain and total score ranges are 0-100, with the higher scores corresponding with better HRQL.
Correlation between FVC measurements and EQ5D | 12 weeks after inclusion
  Correlation between FVC and EQ5D. The EQ5D is a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
Correlation between FVC measurements and EQ5D | 24 weeks after inclusion
  Correlation between FVC and EQ5D. The EQ5D is a standardized instrument to measure health outcomes in two components: health description and valuation. It comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a 5-point scale. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better QoL. In the valuation part the patients' general health status is evaluated using a VAS-score from 0 to 100, with a higher score representing a better QoL.
Correlation between FVC measurements and HADS | 12 weeks after inclusion
  Correlation between FVC and HADS. The HADS is a 14-item questionnaire with 7 questions in the domain anxiety and 7 questions in the domain depression on a 0-3 Likert scale. Higher values represent higher anxiety and depression levels, with a maximum of 21 point in both domains. There is a cut-off score of 8/21 for anxiety and depression.
Correlation between FVC measurements and HADS | 24 weeks after inclusion
  Correlation between FVC and HADS. The HADS is a 14-item questionnaire with 7 questions in the domain anxiety and 7 questions in the domain depression on a 0-3 Likert scale. Higher values represent higher anxiety and depression levels, with a maximum of 21 point in both domains. There is a cut-off score of 8/21 for anxiety and depression.
Correlation between FVC measurements and GRC | 12 weeks after inclusion
  Correlation between FVC and GRC. The Global Rating of Change (GRC) measures whether QoL has improved or deteriorated over a certain period of time, with scores range from -7 to +7, with positive scores corresponding with improvement in QoL.
Correlation between FVC measurements and GRC | 24 weeks after inclusion
  Correlation between FVC and GRC. The Global Rating of Change (GRC) measures whether QoL has improved or deteriorated over a certain period of time, with scores range from -7 to +7, with positive scores corresponding with improvement in QoL.
Correlation between VAS score on stability of IPF scored by patients and healthcare providers | Baseline
  Both patients and healthcare providers will score a Visual Analogue Scale (VAS) with a score between 0 (not stable) and 10 (very stable) on stability of IPF at baseline. Correlation between the VAS scores from patients and healthcare providers will be assessed.
Correlation between VAS score on stability of IPF scored by patients and healthcare providers | 12 weeks
  Both patients and healthcare providers will score the stability of their IPF on a Visual Analogue Scale (VAS). The visual analogue scale has a score between 0 (very unstable) and 10 (very stable), therefore higher scores correspond with better outcomes. Correlation between the VAS scores from patients and healthcare providers will be assessed at 12 weeks.
Correlation between VAS score on stability of IPF scored by patients and healthcare providers | 24 weeks
  Both patients and healthcare providers will score the stability of their IPF on a Visual Analogue Scale (VAS). The visual analogue scale has a score between 0 (very unstable) and 10 (very stable), therefore higher scores correspond with better outcomes. Correlation between the VAS scores from patients and healthcare providers will be assessed at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Wijsenbeek, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moor CC, Mostard RLM, Grutters JC, Bresser P, Aerts JGJV, Dirksen CD, Kimman ML, Wijsenbeek MS. Patient expectations, experiences and satisfaction with nintedanib and pirfenidone in idiopathic pulmonary fibrosis: a quantitative study. Respir Res. 2020 Jul 23;21(1):196. doi: 10.1186/s12931-020-01458-1. PMID 32703201
- [Derived] Moor CC, Mostard RLM, Grutters JC, Bresser P, Aerts JGJV, Chavannes NH, Wijsenbeek MS. Home Monitoring in Patients with Idiopathic Pulmonary Fibrosis. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2020 Aug 1;202(3):393-401. doi: 10.1164/rccm.202002-0328OC. PMID 32325005